CLINICAL TRIAL: NCT03587896
Title: Refugee Emergency: DEFining and Implementing Novel Evidence-based Psychosocial Interventions - The Turkey Site
Brief Title: Implementation of Self Help Plus in Adult Syrian Refugees in Turkey (RE-DEFINE)
Acronym: RE-DEFINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 12-month assessment process has been stopped prematurely due to logistic reasons.
Sponsor: Istanbul Sehir University (Other)
Collaborators: World Health Organization (Other); Universita di Verona (Other)
Responsible Party: Principal Investigator, Ceren Acarturk, Principal Investigator, Istanbul Sehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 779255
Record Dates: First submitted 2018-06-22; First posted 2018-07-16 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Stress; Psychological Distress
Keywords: distress; post-traumatic stress disorder; prevention; refugees; Self Help Plus; Turkey
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: RE-DEFINE is a prospective, randomized, parallel-group trial that will follow study participants over a period of 12-months. Syrian refugees with psychological distress, but without a mental disorder according to the MINI International Neuropsychiatric Interview (M.I.N.I.) for DSM-V and ICD-10, will be randomly assigned to the Self Help Plus intervention or to enhanced treatment as usual (ETAU).
Who Masked: Outcomes Assessor
Masking Description: Participants, facilitators, and research staff involved in the screening and baseline assessment will not be blind to the interventions provided during the trial. Outcomes assessors will be kept blind to the study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self Help Plus (Experimental): SH+ programme has been developed by WHO and collaborators working in the humanitarian field, with expertise in global mental health and psychosocial interventions. SH+ programme consists of a pre-recorded audio course, complemented with bibliotherapy, and thanks to this format not requiring much time from experts for implementation. SH+ consists of 5 sessions.
  Interventions: Behavioral: Self Help Plus
- Enhanced Treatment As Usual (No Intervention): Control arm participants will receive routine social support and/or care according to ordinary practice and following local regulations. Additionally, they will receive baseline and follow-up assessments according to the study schedule, and information about freely available mental health services, social services and community networks providing support to asylum seekers and refugees, and NGOs' contact details.

INTERVENTIONS:
Behavioral: Self Help Plus — 5-session psychosocial intervention
  Arms: Self Help Plus

SUMMARY:
This study evaluates the effectiveness and cost-effectiveness of the SH+ in Arabic speaking people including Syrians under the temporary protection of Republic of Turkey and other Arabic speaking immigrants and asylum seekers with psychological distress in Turkey. Half of participants will receive Self Help Plus (SH+), while the other half will receive enhanced treatment as usual.

DETAILED DESCRIPTION:
Background: Since the start of the war in Syria in 2011, more than 5 million Syrians had to take refuge in a safer place and they had chosen neighbouring countries including Turkey, Lebanon, Jordan, Iraq and countries in Africa including Egypt and North Africa. As a consequence of several adversities, refugees are at great risk of developing symptoms of common mental disorders, notably posttraumatic stress disorder (PTSD), depression, anxiety and related somatic health symptoms along with other forms of disabling psychological distress. The World Health Organization (WHO) has developed a new low-intensity 5-session self-help intervention called Self-Help Plus (SH+) in order to manage stress and cope with adversity (Epping-Jordan et al., 2016). SH+ is a brief and trans-diagnostic intervention which may be delivered by trained non-specialists facilitators to people with and without mental disorders. SH+ has been evaluated in RCTs in low and middle income countries.

Objectives: To evaluate the effectiveness and cost-effectiveness of the Self Help Plus in Arabic speaking people including Syrians under the temporary protection of Republic of Turkey and other Arabic speaking immigrants and asylum seekers with psychological distress resettled in Turkey, as compared with enhanced treatment as usual (ETAU). The primary outcome is the reduction in the incidence of any mental disorders. Secondary outcomes are mental health symptoms, psychological functioning, well-being, drop-out rates, and economic outcomes.

Design: This is a parallel-group randomized controlled trial, in which participants will have an equal probability (1:1) of being randomly allocated to the SH+ intervention or the ETAU.

Methodology: Refugees who screen positive at the General Health Questionnaire (≥ 3) and without a formal diagnosis of any psychiatric disorders according to the M.I.N.I. International Neuropsychiatric Interview (M.I.N.I.) will enter the study. After random allocation they will receive the 5- session SH+ or the ETAU. Assessments will be performed by masked members of the research team immediately after intervention, at 6 months (primary outcome), and a 12 months after randomization.

Time frame: The recruitment phase will last 12 months. After the screening, eligible participants will be assessed at baseline before randomization, immediately post-intervention, and at 6- and 12-month follow-up. The SH+ intervention delivery will be conducted in around 5 weeks (1 session per week).

Expected outcomes: The expected outcomes are a reduction in the incidence of psychiatric diagnoses at 6-month follow-up, and a general improvement in mental health symptoms, psychological functioning, well-being, and economic outcomes at each assessment, in refugees in the SH+ intervention arm, as compared to ETAU.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Able to speak and understand Arabic
* Syrian under temporary protection status
* Presence of psychological distress, as shown by a score of 3 or more at the 12 item General Health Questionnaire (GHQ-12 ≥ 3)

Exclusion Criteria:

* Presence of any mental disorders according to DSM-V and ICD-10, as shown by a positive M.I.N.I.
* Acute medical conditions contraindicating study participation, based on clinical judgment of the health care professional with a clinical background who performs the screening
* Clinical evidence of imminent suicide risk or suicide risk scored as "moderate or high" (or a positive suicidality behaviour disorder) by the M.I.N.I. (section SUICIDALITY)
* Clinical evidence that the decision-making capacity is impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 642 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Psychiatric diagnosis at 6-month follow-up | 6-month follow-up
  The primary outcome will be the number of participants with a current psychiatric diagnosis 6 at six-month follow-up, as measured by the M.I.N.I. The M.I.N.I. was designed as a brief structured interview for the major psychiatric disorders (i.e., major depressive disorder, suicide behavior disorder, post-traumatic stress disorder, social anxiety disorder, etc.) in DSM-5 and ICD-10. The M.I.N.I. is divided into modules identified by letters, each corresponding to a diagnostic category. At the beginning of each module (except for psychotic disorders module), screening question(s) corresponding to the main criteria of the disorder are presented in a gray box. At the end of each module, diagnostic box(es) permit(s) the health care professional to indicate whether the diagnostic criteria are met.

SECONDARY OUTCOMES:
Psychological distress | 1-week post-intervention; 6-month and 12-month follow-ups
  Psychological distress will be measured through the General Health Questionnaire-12. The questionnaire asks whether the respondent has experienced a particular symptom or behaviour recently. Each item is rated on a four-point Likert scale (less than usual, no more than usual, rather more than usual, or much more than usual); and gives a total score of 36 or 12 based on the GHQ version and on the selected scoring methods. Higher scores indicate higher levels of mental distress.
Psychiatric diagnosis | 1-week post-intervention; 6-month and 12-month follow-ups
  Number of participants with a current psychiatric diagnosis as measured by the M.I.N.I.
Functioning | 1-week post-intervention; 6-month and 12-month follow-ups
  The WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) is a generic assessment instrument assessing health and disability. It is used across all diseases, including mental, neurological and substance use disorders. It is simple to administer and applicable across cultures. WHODAS covers six domains (cognition, mobility, self-care, getting along, life activities, and participation). It assesses difficulties people have across these domains during the last 30 days. Difficulties are scored as none, mild, moderate, severe, or extreme. Higher scores indicate higher levels of disability. In the current study, 12-item interviewer-administered version will be used. Data on socio-demographic information (sex, age, education, marital status and work status) will be collected through questions A1-A5 of the WHODAS 2.0, which will be administered first.
Depressive symptoms | 1-week post-intervention; 6-month and 12-month follow-ups
  Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item instrument measuring the presence and severity of depression. Major depression is diagnosed if five or more of the nine depressive symptom criteria have been present at least "more than half the days" in the past two weeks, and one of the symptoms includes depressed mood or anhedonia. Other types of depression are diagnosed if two, three, or four depressive symptoms have been present at least "more than half the days" in the past two weeks, and one of the symptoms includes depressed mood or anhedonia. As a severity measure, the PHQ-9 score may range from 0 to 27, since each of the nine items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores indicate worse symptomatology. The PHQ has been validated for a wide range of cultural groups.
Subjective wellbeing | 1-week post-intervention; 6-month and 12-month follow-ups
  WHO-5 Wellbeing index. The WHO-5 Wellbeing Index is a 5-item questionnaire measuring current psychological wellbeing and quality of life, rather than psychopathology. Each of the items is rated on a 6-point Likert scale from 0 (= not present) to 5 (= constantly present). Scores are summed up and raw scores range from 0 to 25. Then the raw scores are multiplied by 4 and transformed to 0-100. Higher scores indicate better well-being.The scale has demonstrated sensitivity to change in wellbeing and is available in numerous languages.
Self-defined psychosocial goals | 1-week post-intervention; 6-month and 12-month follow-ups
  The Psychological Outcome Profiles instrument (PSYCHLOPS) consists of four questions. It contains three domains: problems (2 questions), function (1 question) and wellbeing (1 question). Participants are asked to give free text responses to the problem and function domains. Responses are scored on an ordinal six-point scale ranging from zero to five, producing a maximum score of 20. Lower scores indicate a better outcome.
Symptoms of post-traumatic stress disorder | 1-week post-intervention; 6-month and 12-month follow-ups
  PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. It takes approximately 5-10 minutes to complete. The PCL-5 can be scored in different ways: (a) a total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items; (b) DSM-5 symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster; (c) a provisional PTSD diagnosis can be made by treating each item rated as 2 = "moderately" or higher as a symptom endorsed, then following the DSM-5 diagnostic rule which requires at least: 1 B item (questions 1-5), 1 C item (questions 6-7), 2 D items (questions 8-14), 2 E items (questions 15-20). Higher scores indicate worse symptomatology. An adapted version making reference to the past week instead of the past month will be used in the current study for sensitivity reasons.
Health-related quality of life | 6-month and 12-month follow-ups
  The EuroQol-5 Dimension-3 level version (EQ-5D-3L). The EQ-5D-3L is applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status that can be used in the clinical and economic evaluation of health care as well as in population health surveys.The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results into a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Cost-effectiveness | 6-month and 12-month follow-ups
  The Client Service Receipt Inventory (CSSRI): Client sociodemographic and service receipt inventory. The CSSRI is a research tool developed for collecting information that describes in detail the types and level of services that comprise the care package of each study member.
Proportion of participants leaving the study early | 12-month follow-up
  Proportion of people leaving the study prematurely at any times, and reasons for discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Ceren Acartürk, Assoc. Prof., Principal Investigator — Koç University
Locations (1):
- Turkish Red Crescent, Mardin, Yenişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epping-Jordan JE, Harris R, Brown FL, Carswell K, Foley C, Garcia-Moreno C, Kogan C, van Ommeren M. Self-Help Plus (SH+): a new WHO stress management package. World Psychiatry. 2016 Oct;15(3):295-296. doi: 10.1002/wps.20355. No abstract available. PMID 27717271
- [Derived] Purgato M, Carswell K, Acarturk C, Au T, Akbai S, Anttila M, Baumgartner J, Bailey D, Biondi M, Bird M, Churchill R, Eskici S, Hansen LJ, Heron P, Ilkkursun Z, Kilian R, Koesters M, Lantta T, Nose M, Ostuzzi G, Papola D, Popa M, Sijbrandij M, Tarsitani L, Tedeschi F, Turrini G, Uygun E, Valimaki MA, Wancata J, White R, Zanini E, Cuijpers P, Barbui C, Van Ommeren M. Effectiveness and cost-effectiveness of Self-Help Plus (SH+) for preventing mental disorders in refugees and asylum seekers in Europe and Turkey: study protocols for two randomised controlled trials. BMJ Open. 2019 May 14;9(5):e030259. doi: 10.1136/bmjopen-2019-030259. PMID 31092670

DOCUMENTS (1):
  • Study Protocol (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03587896/Prot_000.pdf